CLINICAL TRIAL: NCT05262231
Title: The Effect of Online Breastfeeding Education on Breastfeeding Motivation
Brief Title: Online Education and Breastfeeding Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sevgi Özkan, Prof. Dr., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-60116787-020-137020
Record Dates: First submitted 2022-02-12; First posted 2022-03-02 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Birth, First; Breast Feeding; Motivation
Keywords: Breastfeeding motivation; Breastfeeding; Online education; Postpartum period
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Masking Description: The women in the experimental and control groups were not informed about the group they belonged to. However, the researcher had information about the groups in which women were included. In this way, unilateral blinding was achieved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Study group intervention consists 1-session. A session takes approximately 1 hour. The pre-test will be applied just before the intervention. The final test will be administered immediately after the intervention.
  Interventions: Behavioral: Online Breastfeeding Education
- No Intervention (No Intervention): No intervention is applied to the control group.

INTERVENTIONS:
Behavioral: Online Breastfeeding Education — Breastfeeding education will be announced with a poster on social media. At the same time, mothers will be informed about the training in the institution where the institution permission is obtained. Postpartum period 4-8. A single-blind randomization method will be used per week. Pre-test will be applied to the mothers in the experimental and control groups. After the pre-test, online breastfeeding training will be given to the experimental group. The training consists of a single session. It will take about 40-60 minutes. The content of the training includes the benefits of breastfeeding for the mother, baby and society, breast problems and solutions, causes and solutions of breast rejection, breastfeeding positions, etc. consists of topics. After the training experimental group, the post-test will be applied. At the same time, the post-test will be applied to the control group who did not receive the training.
  Arms: Experimental

SUMMARY:
Introduction: Breastfeeding is not just a physiological event. Psychological and emotional factors affect breastfeeding. Motivation is also among these factors. For this reason, it should be considered that there will be problems with breastfeeding in the postpartum period. Since breastfeeding education can be a solution to these problems, it can increase the motivation of mothers for breastfeeding.

Purpose: To examine the effect of online breastfeeding education on breastfeeding motivation.

Methods: The type of the study was planned as a prospective, randomized controlled experimental study with pretest-posttest control group. The sample group of the research will be reached at Pamukkale University Obstetrics and Gynecology clinic and online via social media. The sample reached will be trained in the online environment. The research will be carried out between February 2022 and December 2022. A total of 50 people, 25 in the experimental group and 25 in the control group, will be included. Evaluation will be made with the Breastfeeding motivation scale (for primiparous mothers). Motivation scores will be compared before and after the training.

DETAILED DESCRIPTION:
Breastfeeding protects children against diseases such as gastrointestinal, asthma, diabetes, otitis media, sudden infant death syndrome and obesity. At the same time, it supports the increase of children's IQ level and brain development. Among the benefits for women's health are its contribution to the involution process in the postpartum period, protection against postpartum depression, ovarian and breast cancer. The social impact of breastfeeding is that it provides economic benefits.Despite all the benefits of breastfeeding, breastfeeding rates are not sufficient. Globally, the rate of exclusive breastfeeding of children for the first six months is 41%, and the rate of breastfeeding with complementary foods for two years is 45%.

There are many factors that affect breastfeeding. These; social, environmental, cultural and personal factors. These factors can affect the motivation of women internally and externally.For this reason, internal and external motivations of women will be supported with breastfeeding education.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-49 years old,
* Having given birth for the first time,
* Being in the postpartum period between the 4th and 8th weeks and breastfeeding,
* Volunteering to participate in the research,
* Speak and understand Turkish.

Exclusion Criteria:

* not be between the ages of 18-49,
* Having more than one birth,
* not breastfeeding,
* Not being able to speak or understand Turkish.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Yes
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Motivation Scale (For Primiparous Mothers) | Change in motivation after a one-session training of approximately 1 hour
  The breastfeeding motivation scale developed for primiparous women consists of 23 questions.Intrinsic motivation consists of five sub-factors: integrated regulation, identified regulation, introjected regulation, and extrinsic regulation.The scale, which is a four-point Likert type scale, is scored as 1 = I strongly disagree, 2 = I do not agree, 3 = I agree, 4 = I strongly agree. Total points are not taken from the scale. As the score obtained from the scale sub-dimension increases, the motivation representing that sub-dimension also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

REFERENCES:
- [Result] Cangol E, Sahin NH. The Effect of a Breastfeeding Motivation Program Maintained During Pregnancy on Supporting Breastfeeding: A Randomized Controlled Trial. Breastfeed Med. 2017 May;12:218-226. doi: 10.1089/bfm.2016.0190. Epub 2017 Mar 13. PMID 28287819
- [Result] Khasawneh W, Kheirallah K, Mazin M, Abdulnabi S. Knowledge, attitude, motivation and planning of breastfeeding: a cross-sectional study among Jordanian women. Int Breastfeed J. 2020 Jul 1;15(1):60. doi: 10.1186/s13006-020-00303-x. PMID 32611353
- [Result] Louis-Jacques AF, Stuebe AM. Enabling Breastfeeding to Support Lifelong Health for Mother and Child. Obstet Gynecol Clin North Am. 2020 Sep;47(3):363-381. doi: 10.1016/j.ogc.2020.04.001. Epub 2020 Jul 2. PMID 32762923
- [Result] Peven K, Purssell E, Taylor C, Bick D, Lopez VK. Breastfeeding support in low and middle-income countries: Secondary analysis of national survey data. Midwifery. 2020 Mar;82:102601. doi: 10.1016/j.midw.2019.102601. Epub 2019 Dec 10. PMID 31935650
- [Derived] Yildirim Goksen DF, Ozkan S. The effect of online breastfeeding education on breastfeeding motivation: A randomized controlled study. J Pediatr Nurs. 2024 Mar-Apr;75:e42-e48. doi: 10.1016/j.pedn.2023.12.026. Epub 2024 Jan 5. PMID 38182483